CLINICAL TRIAL: NCT05783674
Title: The Effect of Physical Activity and Exercise by Brain Breaks®️ Video Games on Sleep and Life Quality of People With Mental Health Problems
Brief Title: The Effect of Brain Breaks on People With Mental Health Problems
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istinye University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2239
Record Dates: First submitted 2023-03-14; First posted 2023-03-24 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Physical Inactivity
Keywords: Mental Health Problems; BrainBreaks; Sleep Quality; Quality of Health
MeSH Terms: conditions — Sedentary Behavior; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BrainBreaks for people without mental health problems (Experimental): BrainBreaks for people without mental health problems
  Interventions: Other: Brain Breaks® Video Exercises; Other: Posture training
- BrainBreaks for people with mental health problems (Experimental): BrainBreaks for people with mental health problems
  Interventions: Other: Brain Breaks® Video Exercises; Other: Posture training

INTERVENTIONS:
Other: Brain Breaks® Video Exercises — A total of at least 140 Brain Breaks® videos, each 3-4 minutes long, aerobic exercises including wide joint movements, movements specific to different sports branches such as yoga and volleyball, basketball, football, tennis, karate, judo, and warm-up-cooling movements. It includes national dances of different cultures. Horon, Zeybek, Scarf dance, morning gymnastics in Ürgüp Göreme, dribbling (volleyball, basketball), Pilates ball, and core area exercises. In each session, 2 videos will be applied and each will be repeated 2-3 times, and a 3-minute rest break will be given between each video. The total session will last for 20-30 minutes on average and physical activity will be performed twice a week, for a total of 8 weeks, 16 sessions.
Other: Posture training — All participants, as the BB Video Exercise and Control Group, will be given a 20-minute hands-on training on the importance of proper posture once at the beginning of the study, and breathing control training will be given to maintain proper sitting, standing, lying postures, and proper posture.

SUMMARY:
Regular physical activity (PA) and adopting an active lifestyle protect against non-communicable diseases such as diabetes, cardiovascular diseases, hypertension, obesity, and colon cancer in the general population. However, the habit of doing regular FA in societies is quite low. It is reported that those adopting a sedentary lifestyle in the general population range from 16.3% to 39.1%, with an average of 27.5%. These values indicate that the risk of contracting non-communicable diseases can be reduced by developing the habit of doing FA for almost one-third of the population. Based on this idea, the World Health Organization has decided to increase FA by 10% among the "Nine Global Goals" it has addressed against the spread of non-communicable diseases.

People with mental health problems are less active than the general population. For example, it is reported that people diagnosed with major depression syndrome are 50% less active than their peers. Dikerson et al. reported that people with mental illnesses are 50% more obese than their peers. Verhoeven et al. They concluded that people with severe and chronic depression will age biologically earlier (7-10 years) than their peers. They emphasized the importance of lifestyle changes in the prevention of biological aging and possible diseases (coronary diseases, type-2 diabetes, obesity, dementia, cancer).

Marquez et al. also indicate that there is a significant relationship between mental illnesses and chronic medical problems such as cancer, cardiovascular diseases, diabetes, and obesity. Therefore, increasing the habit of regular PA and exercise among people with mental health problems is important in protecting against diseases. Our study aims to adopt the habit of doing physical activity accompanied by technology-supported GCH Brain Breaks®️ videos applied to people with mental health problems; In this context, at least 20 minutes of video-accompanied FA and exercise and 30 minutes of exercise in individuals every day to gain the habit of walking.

DETAILED DESCRIPTION:
The fact that the group addressed by our study is unique and that these entertaining video exercises have not been previously applied to adults and people with mental health problems makes our study unique. At the same time, we believe that the level of physical activity increased by technology-supported HOPSports Brain Breaks® videos applied to people with mental health problems will improve sleep quality, general physical condition, and life satisfaction of people. This result, which we plan to reach, also increases the originality of our study. Therefore, it is expected that the functional and social results of our technology-assisted FA and exercise program, which will be given to people with mental problems, will contribute to the national and international literature.

Therefore, our study aims to adopt the habit of doing physical activity accompanied by technology-supported GCH Brain Breaks®️ videos applied to people with mental health problems; In this context, at least 20 minutes of video-accompanied FA and exercise and 30 minutes of exercise in individuals every day. to gain the habit of walking.

ELIGIBILITY:
Inclusion Criteria:

* To be diagnosed with one of the mental health problems,
* Being over 25 years old and male,
* T.C. Being a resident of Istanbul Governorship Beylikdüzü Disabled Life Care, Rehabilitation and Family Counseling Center or Carnation Care Center located in Kemerburgaz Büyükçekmece,
* To volunteer to participate in the study

Exclusion Criteria:

* Having a serious chronic illness,
* It is a notification that physical activity and exercise are not appropriate due to a serious mental illness.

Ages: 25 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Due to hormonal levels the study will be done on a single sex.
Enrollment: 52 (Estimated)
Dates: Start 2023-03-05 (Actual); Primary Completion 2023-05-03 (Estimated); Study Completion 2023-06-03 (Estimated)

PRIMARY OUTCOMES:
pittsburgh sleep quality index | 12 weeks
  Sleep quality will be evaluated with the Pittsburg Sleep Quality Index (PUKI), developed by Buysse et al. (1989) and adapted into Turkish by Ağargün et al. (1996). PUKI is a 19-item self-report scale that evaluates sleep quality and disturbance in the past month. It consists of 24 questions, 19 questions are self-report questions, and 5 questions are questions to be answered by the spouse or roommate.
Contentment with Life Scale | 12 weeks
  The Content with Life Scale, consisting of 5 items, developed by Lavallee et al. (2007) will be used to evaluate life satisfaction. This one-dimensional scale has a 7-point Likert-type rating ("1" strongly disagree- "7" strongly agree).

SECONDARY OUTCOMES:
6 minutes walking test | 12 weeks
  The six-minute walk test (6 MWT) is the most commonly used submaximal exercise test in clinical practice. In a long corridor (30 meters), the patient is asked to walk at normal walking speed for 6 minutes. The time will be measured with a stopwatch. It is calculated how many meters the patient has traveled after the test.
Visual Pain Scale | 12 weeks
  It is a frequently used evaluation method to convert the severity of pain that cannot be measured numerically into numerical data. Above a 100mm line, the person marks where he or she describes his condition. The far left of the line is defined as "I have no pain" and the far right is defined as "I have very severe pain". Data is obtained by measuring the distance between the place marked by the patient and the place where he has no pain.
New York Posture Assessment Test | 12 weeks
  Postures of individuals were determined by the New York Posture Assessment Test, thirteen (13) regions of the body from the back (head-A, shoulder levels-B, vertebral column-C, hip levels-D, mediolateral position of the feet-E, foot arches-F) and side ( head-G, rib cage-H, shoulders-I, upper back-J, trunk-K, abdomen-L, lower back-waist-M) will be observed and scored on the form.
268 / 5.000 Çeviri sonuçları Çeviri sonucu Muscle Elasticity | 12 weeks
  Shortness-Flexibility assessment Hamstrings, Lumbal extensors, Pectorals, Tensor Fascia Latae, and Gastrocnemius muscles (short:3, moderately short:2, and normal:1) will be evaluated. Measurements will be made separately for the right and left sides of the body.
Muscle Strength | 12 weeks
  As peripheral muscle strength, quadriceps femoris, tibialis anterior, tibialis posterior, extensor hallucis, flexor hallucis, gastrocnemius, soleus, hamstring gluteus maximus, gluteus medius, back extensor muscles, abdominal muscles strength, portable manual muscle strength measuring device myometer (Model 01165, IN, USA) in kg. Measurements for the right and left sides will be repeated three times and the best value obtained will be recorded in Newtons (N). Measurements 15 min. is expected to last.
Body Mass Index | 12 weeks
  The main variables to be used as a reference in anthropometric evaluations, body mass index, were preferred especially because it is an easy and fast measurement method in the clinic and a primary obesity assessment tool for adults. BMI data of individuals will be calculated by dividing the body weight in kilograms by the square of the height in meters.

CONTACTS AND LOCATIONS:
Locations (1):
- Istinye University, Istanbul, Zeytinburnu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No